CLINICAL TRIAL: NCT01212562
Title: Open Label, Phase 3 Study of the Efficacy of Combination of Imiquimod and Cryosurgery in the Treatment of Primary Basal Cell Carcinomas of the Skin
Brief Title: Treatment of Primary Basal Cell Carcinomas of the Skin With Combination of Topical Imiquimod and Cryosurgery
Acronym: IMCX
Status: Completed | Type: Observational
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Ioannis Bassukas, Associate Professor of Dermatology, University of Ioannina
Other Study IDs: 75090409
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Basal Cell Carcinoma
Keywords: basal cell carcinoma; cryosurgery; imiquimod; immunocryosurgery
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Imiquimod

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples with anticoagulant at -20C
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Immunocryosurgery: 2 weeks daily imiquimod application prior to a session of cryosurgery and subsequently 3 weeks continued daily imiquimod application
  Interventions: Procedure: Immunocryosurgery

INTERVENTIONS:
Procedure: Immunocryosurgery — Assessing the efficacy of cryosurgery during continued imiquimod application (immunocrysurgery) in the treatment of basal cell carcinoma of the skin
  Other Names: Aldara

SUMMARY:
The purpose of this study is to evaluate the efficacy of cryosurgery during continuing imiquimod application in the treatment of basal cell carcinoma of the skin.

DETAILED DESCRIPTION:
Evaluation of efficacy:

* Number of patient: N=50
* Inclusion criteria: Basal cell carcinoma of the skin proven with biopsy
* Exclusion criteria: (1) Size of the tumors >2cm; (2) Distance from the eyelid <1cm; (3)Number of tumors >5

Treatment protocol: Patients will apply imiquimod daily for 14 days on the tumor and a rim of 2mm around the tumor. On day 14 a session of mild cryosurgery (2 cycles of 10-15 seconds, with open spray liquid nitrogen) will be applied and the patients will continue application of imiquimod for another 3 weeks before being evaluated again. Persisting erosion will be considered as persistence of the tumor and imiquimod will be continued for another 3 weeks with/or without a cryosurgery session. The patients will be evaluated at 1,3,6,12 months after discontinuation of imiquimod and yearly thereafter for relapse. In case of clinical relapse, it will be confirmed by biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Basal cell carcinoma of the skin
* Size < or = 2cm
* Number of tumors < or = 5
* Distance from eyelids, mouth >1cm

Exclusion Criteria:

* Size >2cm Number of tumors > 5 Distance from eyelids or mouth < or = 1cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with basal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of immunocryosurgery in the treatment of basal cell carcinoma of the skin | 1 months
  Basal cell carcinomas of the skin will be treated with immunocryosurgery and the efficacy will be measured 1, 3, 6, and 12 months. Reappearance of the tumor within the primary lesion and 1cm around it will be considered as relapse.

SECONDARY OUTCOMES:
Feasibility and Tolerability of Immunocryosurgery | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis D Bassukas, Professor, Principal Investigator — Medical School, University of Ioannina
Locations (1):
- Department for Skin and Venereal Diseases, University Hospital, Ioannina, Greece

REFERENCES:
- [Background] Bassukas ID, Gaitanis G. Combination of cryosurgery and topical imiquimod: does timing matter for successful immunocryosurgery? Cryobiology. 2009 Aug;59(1):116-7. doi: 10.1016/j.cryobiol.2009.04.011. Epub 2009 May 6. No abstract available. PMID 19426725
- [Background] Bassukas ID, Gamvroulia C, Zioga A, Nomikos K, Fotika C. Cryosurgery during topical imiquimod: a successful combination modality for lentigo maligna. Int J Dermatol. 2008 May;47(5):519-21. doi: 10.1111/j.1365-4632.2008.03562.x. PMID 18412875
- [Background] Gaitanis G, Mitsou G, Tsiouri G, Alexis I, Bassukas ID. Cryosurgery during imiquimod cream treatment ("immunocryosurgery") for Bowen's disease of the skin: a case series. Acta Derm Venereol. 2010 Sep;90(5):533-4. doi: 10.2340/00015555-0896. No abstract available. PMID 20814639
- [Result] Gaitanis G, Nomikos K, Vava E, Alexopoulos EC, Bassukas ID. Immunocryosurgery for basal cell carcinoma: results of a pilot, prospective, open-label study of cryosurgery during continued imiquimod application. J Eur Acad Dermatol Venereol. 2009 Dec;23(12):1427-31. doi: 10.1111/j.1468-3083.2009.03224.x. Epub 2009 Jun 25. PMID 19555364
- [Derived] Gaitanis G, Bassukas ID. Immunocryosurgery for non-superficial basal cell carcinomas </= 20 mm in maximal diameter: Five-year follow-up. J Geriatr Oncol. 2019 May;10(3):475-478. doi: 10.1016/j.jgo.2018.08.012. Epub 2018 Sep 12. PMID 30219274